CLINICAL TRIAL: NCT06234501
Title: Testing the Potential of High-dose Vitamin B6 Supplements for Sensory Reactivity in Autism
Brief Title: Testing the Efficacy of 100mg Vitamin-B6 Daily for Sensory Reactivity in Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: INNOPURE (Unknown)
Responsible Party: Principal Investigator, David Field, Associate professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UREC23/27
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Autism
Keywords: Vitamin B6; Sensory Hyperreactivity; GABA; Excitation-Inhibition Balance
MeSH Terms: conditions — Autistic Disorder | interventions — Pyridoxal Phosphate; Vitamin B 6; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin-B6 (Experimental): Participants will consume one high-dose Vitamin B6 100 mg tablet orally once daily for one month. Vitamin B6 will be provided as Pyridoxal-5'-Phosphate (PLP)
  Interventions: Dietary Supplement: Pyridoxal 5'-Phosphate (100 mg)
- Placebo (Placebo Comparator): Participants will consume a Placebo tablet matching the appearance of the Vitamin B6 tablets in the Experimental arm orally once daily for one month.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pyridoxal 5'-Phosphate (100 mg) — 100 mg Pyridoxal 5'-Phosphate tablet once daily with food
  Other Names: Vitamin B6
  Arms: Vitamin-B6
Other: Placebo — Placebo tablet once daily
  Other Names: Control group
  Arms: Placebo

SUMMARY:
This clinical trial aims to explore the effect of Vitamin B6 supplementation on anxiety sensory hyperreactivity in autistic adults. Researchers will compare a placebo group to high-dose Vitamin-B6 to see if vitamin B6 reduce anxiety and sensory reactivity differences in autism.

DETAILED DESCRIPTION:
The main question it aims to answer is:

* Does high-dose Vitamin B6 supplementation reduce sensory hyperreactivity differences in autism?
* Does high-dose Vitamin B6 supplementation reduce anxiety differences in autism?
* Explore the effects of vitamin B6 on sleep quality, Attention Deficit Hyperactivity Disorder (ADHD) scores, and various visual perception tasks that are indicative of GABAergic activity

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 60
* With a diagnosis of autism

Exclusion Criteria:

* Taking any supplement that contains more than 2mg of Vitamin B6 or taking GABA agonist drugs
* Have a medical history of peripheral neuropathy
* lactose intolerance (placebo tablet is lactose based)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Sensory hyperreactivity | Baseline and One month
  Sensory hyperreactivity will be measured by a subscale of the Sensory Processing Inventory (SP3D.
Sensory hyperreactivity | Baseline and One month
  Sensory hyperreactivity will be measured by a subscale of the Comprehensive Autistic Trait Inventory (CATI).
Anxiety | Baseline and One month
  Anxiety will be measured using the Screen for Adult Anxiety Related Disorders (SCAARED) questionnaire.
Vitamin B6 status | Baseline and One month
  The concentration of different forms of Vitamin B6 in blood plasma will be measured (Pyridoxal-5'-phosphate, pyridoxine, pyridoxal, pyridoxamine)

SECONDARY OUTCOMES:
ADHD traits | Baseline and One month
  Adult Attention Deficit Hyperreactivity Disorder Self-Report Scale (ASRS-v1.1)
Sensory processing differences | Baseline and One month
  These will be measured using the other subscales of the Sensory Processing Inventory (SP3D) that do not constitute the primary sensory hyperreactivity outcome described above.
Sleep quality | Baseline and One month
  Pittsburgh Sleep Quality Index (PSQI)
Visual Surround Suppression of contrast perception | Baseline and One month
  Psychophysical measurements of the contrast threshold will be made, which correspond to the minimum physical stimulus contrast that can be reliably detected by an observer. The test measures the increase in the threshold caused by introducing spatial inhibition of the target stimuli, which is a parameter that has been shown to correlate with GABA concentration in the brain (Yoon et al., 2010).
Surround Suppression of Motion duration detection thresholds | Baseline and One month
  Psychophysical measurements of the motion duration threshold will be made, which correspond to the number of milliseconds an observer requires to detect whether a Gabor patch is drifting left or right. The test measures the increase in the threshold caused by spatial inhibition, which is a parameter that has been shown to differ in various patient groups, including autism (Foss-Feig et al. 2013).
Binocular Rivalry reversal rate | Baseline and One month
  A test based on presenting ambiguous visual stimuli that cause perceptual reversals; how frequently the perceptual reversals occur is measured and has been shown to be related to GABA levels (Mentch et al., 2019).
Binocular Rivalry suppression index | Baseline and One month
  A test based on presenting ambiguous visual stimuli that cause perceptual reversals; the proportion of time for which the stimulus appears unclear rather than stable is measured and has been shown to be related to GABA levels (Mentch et al., 2019).
Measurement of Weber Fraction for size perception | Baseline and One month
  The Weber fraction is the percentage change in a physical quantity required for an observer to reliably detect that a change has occurred, and for a specific stimulus type it is generally a fixed percentage regardless of the magnitude of the stimuli. We will measure the Weber Fraction for visual size perception at four separate starting sizes, and the outcome measure derived from doing that will be a measurement of the stability/instability of the Weber Fraction across the four starting sizes. It has been reported that in autism the general finding of fixed Weber fractions across a range of physical stimuli does not hold (Hadad & Schwartz, 2019): we are taking the opportunity to replicate this finding.
Tilt illusion magnitude | Baseline and One month
  Magnitude of the tilt illusion is a correlate of GABA concentration in the occipital cortex (Song et al., 2017).
Ebbinghaus illusion magnitude | Baseline and One month
  Magnitude of the Ebbinghaus illusion is a correlate of gamma y-Aminobutyric acid (GABA) concentration in the parietal lobe (Song et al. 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Dr David T Field, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon JH, Maddock RJ, Rokem A, Silver MA, Minzenberg MJ, Ragland JD, Carter CS. GABA concentration is reduced in visual cortex in schizophrenia and correlates with orientation-specific surround suppression. J Neurosci. 2010 Mar 10;30(10):3777-81. doi: 10.1523/JNEUROSCI.6158-09.2010. PMID 20220012
- [Background] Mentch J, Spiegel A, Ricciardi C, Robertson CE. GABAergic Inhibition Gates Perceptual Awareness During Binocular Rivalry. J Neurosci. 2019 Oct 16;39(42):8398-8407. doi: 10.1523/JNEUROSCI.0836-19.2019. Epub 2019 Aug 26. PMID 31451579
- [Background] Song C, Sandberg K, Andersen LM, Blicher JU, Rees G. Human Occipital and Parietal GABA Selectively Influence Visual Perception of Orientation and Size. J Neurosci. 2017 Sep 13;37(37):8929-8937. doi: 10.1523/JNEUROSCI.3945-16.2017. Epub 2017 Aug 14. PMID 28821653
- [Background] Hadad BS, Schwartz S. Perception in autism does not adhere to Weber's law. Elife. 2019 Mar 4;8:e42223. doi: 10.7554/eLife.42223. PMID 30829198
- [Background] Foss-Feig JH, Tadin D, Schauder KB, Cascio CJ. A substantial and unexpected enhancement of motion perception in autism. J Neurosci. 2013 May 8;33(19):8243-9. doi: 10.1523/JNEUROSCI.1608-12.2013. PMID 23658163